CLINICAL TRIAL: NCT02861989
Title: Qualitative Study on Representations of Osteoporosis in the General and At-risk Population and in General Practitioners.
Brief Title: Qualitative Study on Osteoporosis Representation and Management in the General Population and in General Practitioners.
Acronym: QUALIOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0499
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Osteoporosis
Keywords: osteoporosis; prevention; care management; focus groups
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Osteoporotic women: women over 50 years with a diagnosis of osteoporosis or history of fragility fracture /osteoporosis treatment
  Interventions: Other: qualitative study
- At risk women: women over 50 years without a diagnosis of osteoporosis or history of fragility fracture /osteoporosis treatment
  Interventions: Other: qualitative study
- Osteoporotic men: Men over 60 years with a diagnosis of osteoporosis or history of fragility fracture /osteoporosis treatment
  Interventions: Other: qualitative study
- At-risk men: Men over 60 years without a diagnosis of osteoporosis or history of fragility fracture /osteoporosis treatment
  Interventions: Other: qualitative study
- General practitioners: General practitioners from the Rhône area, France
  Interventions: Other: qualitative study

INTERVENTIONS:
Other: qualitative study

SUMMARY:
Osteoporosis (OP) and subsequent fractures (OP fractures) are a source of morbidity and high mortality in the elderly. Despite numerous programs aiming at improving OP care, the prevention, diagnostic and treatment remain suboptimal. Barriers to a better care are multiple, both in the general and at-risk population, and in medical practitioners. Since they do not perceive their susceptibility to OP, people do not see the benefit of prevention. In addition, physicians do not give sufficient importance to OP prevention and care, despite the existence of guidelines.

The investigators implemented a qualitative study to explore the knowledge and representations regarding osteoporosis in the general and at-risk population and in doctors in Rhône-Alpes Region, France, using focus groups with women and men and semi-structured face-to-face interviews with general practitioners. Understanding barriers to osteoporosis care in patients and general practitioners will help to set up effective strategies to improve prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* group 1: women aged 50 to 85 years with a history of fragility fracture or an osteoporosis diagnostic
* group 2: women aged 50 to 85 years without a history of fragility fracture or an osteoporosis diagnostic
* group 3: men aged 60 to 85 years with a history of fragility fracture or an osteoporosis diagnostic
* group 4: men aged 60 to 85 years without a history of fragility fracture or an osteoporosis diagnostic
* group 5: general practitioners in Region Rhône-Alpes, France
* who signed the consent form

Exclusion Criteria:

* no signed consent
* legal disability
* difficulty in understanding French
* psychiatric disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women aged 50 to 85 years and men aged 60 to 85 years, and general practitioners.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Focus Group Interview | 24 hours
  Representations of osteoporosis, in general practitioners and in 4 groups of people.
  Representations were drawn from focus groups interviews based on the theory of social representations of illness developed by Moscovici and Durkheim. Four types of focus groups were conducted until data saturation: 9 groups with women aged 50 to 85 years and 7 groups with men aged 60 to 85 years, with or without a history of fragility fracture or an osteoporosis diagnostic.
  In parallel, semi-structured face-to face interviews were conducted with 16 general practitioners

SECONDARY OUTCOMES:
Factors favoring and barriers to a better management of OP in each group | At the day of inclusion
  Factors favoring and barriers to a better management of OP were collected during the focus groups interviews. Specific questions were asked to collect information on reasons for not complying with recommendations or prescriptions. Four types of focus groups were conducted until data saturation: 9 groups with women aged 50 to 85 years and 7 groups with men aged 60 to 85 years, with or without a history of fragility fracture or an osteoporosis diagnostic.
  In parallel, semi-structured face-to face interviews were conducted with 16 general practitioners
Specific communication needs for the different groups: men/women, fractured/non-fractured. | At the day of inclusion
  Needs for communication tools were collected by specific questions asked during the focus groups interviews. Four types of focus groups were conducted until data saturation: 9 groups with women aged 50 to 85 years and 7 groups with men aged 60 to 85 years, with or without a history of fragility fracture or an osteoporosis diagnostic.
  In parallel, semi-structured face-to face interviews were conducted with 16 general practitioners

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Schott, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Pôle IMER, Hospices Civils de Lyon, Lyon, France